CLINICAL TRIAL: NCT01141933
Title: Creating Meaning Following Cancer: An Cognitive-existential Intervention to Improve Existential and Global Quality of Life
Brief Title: Creating Meaning Following Cancer: An Intervention to Improve Existential and Global Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Laval University (Other); Centre de recherche en cancérologie de l'Université Laval (Unknown); Canadian Cancer Society (CCS) (Other); Maison Michel-Sarrazin (Unknown)
Responsible Party: Principal Investigator, Pierre Gagnon, MD, FRCPC, Psychiatrist, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: CSS-019126
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Non-metastatic Cancer; Adjustment Disorder
Keywords: Creating meaning; Therapy; Cancer; Oncology; Existential; Spirituality; Quality of life; QOL; Psycho-oncology; French-canadian; Cognitive therapy; Existentialism
MeSH Terms: conditions — Adjustment Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (Other): Subjects in this group receive the usual treatment only.
  Interventions: Other: Usual care
- Individual intervention (Experimental): Consisting in a 12 weekly sessions with a therapist. Each session lasts 1 hour.
  Interventions: Other: Cognitive-existential intervention
- Group intervention (Experimental): Consisting in a 12 weekly sessions with two therapists. Number of subjects in each group is from 5 to 10. Each session lasts 2 hours.
  Interventions: Other: Cognitive-existential intervention

INTERVENTIONS:
Other: Cognitive-existential intervention — Over the past 2 years we developed a 12-week cognitive-existential intervention consisting of 12 modules. The first three modules essentially involve cognitive and behavioral techniques proposing reinforcement of the use of active behavioral (e.g., relaxation, activation) and emotional (cognitive reframing) strategies. This content comes from classical cognitive-behavioral techniques. The next 3 modules, inspired by empirically-tested interventions further explore emotional strategies. The last six modules specifically address the existential dimension. They are adapted from logotherapy techniques, which are also empirically-based, and have been adapted to a French-Canadian culture by our team. They aim to improve meaning-based and emotional coping strategies.
  Arms: Group intervention; Individual intervention
Other: Usual care — This group receive the usual treatment only.
  Arms: Usual care

SUMMARY:
The purpose of this study is to test the efficacy of a cognitive-existential intervention (using either an individual or a group format) to improve the existential and global quality of life of patients as compared to usual care in a population of adult non-metastatic cancer patients.

DETAILED DESCRIPTION:
People diagnosed with cancer must learn to cope with loss of meaning and empowerment which compromises quality of life. Questions regarding "Why me?", along with universal existential concerns about death, search for meaning, and sense of control over one's life, often constitute the principal source of overall suffering. Since there is no single and identifiable cause for cancer, those existential questions are commonly observed among patients who demand specific interventions to properly address this central issue. The existential approach can be used to help patients find meaning in the midst of a crisis. It addresses a central issue of survivorship in cancer.

The conceptual model explains the relation between being exposed to a stressful and traumatic life event such as cancer and the risk of progressing toward adjustment difficulties which compromises quality of life and existential integrity. Cancer constitutes a major stressor involving significant losses that confronts the person's beliefs system. A set of therapeutic strategies can help to cope with this inevitable challenge: 1) cognitive-behavioral strategies; 2) direct existential intervention; and 3) social support through supportive-expressive strategies. Adjustment first involves cognitive reframing of the perception of the situation (situational meaning). Cognitive reframing also contributes to a readjustment of personal beliefs and values (global meaning and existential dimension). Existential strategies enable to further this process by including cognitive (beliefs, sense of coherence, expectations), motivational (choice, goal setting, and goal driving) and affective dimensions. The expressive-supportive strategy promotes active listening and non-judgmental support to encourage expression of emotions. The use of these active coping strategies (meaning-based) to the threatened-life challenge enables optimization of existential and global quality of life, as opposed to employing passive strategies such as avoidance.

ELIGIBILITY:
Inclusion Criteria:

* Be of 18 years of age or more;
* Speak French;
* Have received a diagnosis of non-metastatic cancer;
* Be available to participate in the program of 12 weekly group or individual sessions.

Exclusion Criteria:

* Depressive mood (score greater than 10 on the Hospital Anxiety and Depression Scale depressive subscale) that could interfere with the intervention. Since we specifically target the existential dimension and it might temporarily provoke questioning in patients, high psychological distress must first be addressed using other approaches.
* Diagnosis of metastatic cancer or diagnosis of non-metastatic cancer with a usually fast-growing and unpredictable course, making it unlikely to adhere to the intervention (e.g., pancreatic cancer, acute leukemia, glioblastoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Estimated)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Existential quality of life | T0: Pre-intervention
  At every time frame, we use two questionnaires to measure the primary outcome:
  1. The McGill Quality of Life Questionnaire (MQOL): 16 items plus a single-item global scale.
  2. Spiritual well-being (FACIT-SP): The FACIT-SP is a sub-scale of the FACT-G (Functional Assessment of Cancer Therapy-General) and a French version of the "FACIT-SP, FACIT-Spiritual well-being scale". This questionnaire has two sub-scales: Meaning/Peace (8 items) and Faith (4 items).
Existential quality of life | T1: Mid-intervention (6 weeks after the beginning of the intervention)
Existential quality of life | T2: End of the intervention (12 weeks after the beginning of the intervention)
Existential quality of life | T3: First follow-up measure (3 months after the end of the intervention)
Existential quality of life | T4: Second follow-up measure (6 months after the end of the intervention)
Existential quality of life | T5: Last follow-up measure (12 months after the end of the intervention)

SECONDARY OUTCOMES:
Global quality of life | T0: Pre-intervention
  To measure the secondary outcome, The McGill Quality of Life Questionnaire (MQOL) is use at every time frames.
Global quality of life | T1: Mid-intervention (6 weeks after the beginning of the intervention)
Global quality of life | T2: End of the intervention (12 weeks after the beginning of the intervention)
Global quality of life | T3: First follow-up measure (3 months after the end of the intervention)
Global quality of life | T4: Second follow-up measure (6 months after the end of the intervention)
Global quality of life | T5: Last follow-up measure (12 months after the end of the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Gagnon, MD, FRCPC, Principal Investigator — Laval University
Locations (5):
- Canada (5):
  - University of Manitoba, Winnipeg, Manitoba
  - Centre hospitalier affilié universitaire de l'Hôtel-Dieu de Lévis, Lévis, Quebec
  - McGill University, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec

REFERENCES:
- [Background] Gagnon, P., Fillion, L., Girard, M.La recherche de sens à la suite d'un diagnostic de cancer: une invervention pour améliorer la qualité de vie existentielle et globale.Les cahiers francophones de soins palliatifs 9 (1): 57-69, 2008.
- [Background] Gagnon P, Fillion L, Robitaille MA, Girard M, Tardif F, Cochrane JP, Le Moignan Moreau J, Breitbart W. A cognitive-existential intervention to improve existential and global quality of life in cancer patients: A pilot study. Palliat Support Care. 2015 Aug;13(4):981-90. doi: 10.1017/S147895151400073X. Epub 2014 Jul 22. PMID 25050872
- See also: Laval University Cancer Research center - Dr Pierre Gagnon — https://www.crc.ulaval.ca/la-recherche/chercheurs-reguliers/fiche/show/gagnon-pierre/